CLINICAL TRIAL: NCT04342013
Title: Impact of a Novel Electronic Clinical Decision Support Application on Perioperative Medication Errors and Adverse Medication Events: a Randomized Controlled Trial
Brief Title: RCT: The Effect of an Electronic Clinical Decision Support Application on Perioperative Medication Errors.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karen C. Nanji,M.D.,M.P.H. (Other)
Responsible Party: Sponsor-Investigator, Karen C. Nanji,M.D.,M.P.H., Assistant Professor of Anesthesia at Harvard Medical School, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K08HS024764 (AHRQ)
Record Dates: First submitted 2020-04-01; First posted 2020-04-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Perioperative Medication Errors; Perioperative Adverse Medication Events
Keywords: medication safety; perioperative; anesthesiology; clinical decision support

STUDY DESIGN:
Intervention Model Description: Randomized, non-blinded, parallel-arm clinical trial to assess the incidence of medication errors and adverse medication events with and without the use of an electronic clinical decision support application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative Clinical Decision Support Application (Experimental): Participants will be observed performing clinical tasks and documenting medication administrations with use of the clinical decision support application in the perioperative setting.
  Interventions: Other: Electronic Clinical Decision Support Application
- No Perioperative Clinical Decision Support Application (No Intervention): Participants will be observed performing clinical tasks and documenting medication administrations without use of the clinical decision support application in the perioperative setting.

INTERVENTIONS:
Other: Electronic Clinical Decision Support Application — Robust, real-time medication-related clinical decision support application for use in the operating room. The application is fully integrated with existing clinical systems. It provides visual alerts for medication errors and adverse medication events at the point-of-care.
  Arms: Perioperative Clinical Decision Support Application

SUMMARY:
The purpose of this study is to assess the effect of a novel clinical decision support application on the rate of perioperative medication errors and preventable adverse medication events. The investigators hypothesize that the perioperative clinical decision support application will reduce the incidence of perioperative medication errors and adverse medication events compared to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia clinician (anesthesiologists, certified registered nurse anesthetists (CRNAs), student nurse anesthetists, fellows and residents) at Massachusetts General Hospital.

Exclusion Criteria:

* Study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Combined incidence of medication errors and adverse medication events in the perioperative setting | 6 months
  Number of medication errors and adverse medication events / number of medications administered

SECONDARY OUTCOMES:
Incidence of medication errors the perioperative setting | 6 months
  Number of errors / number of medications administered
Incidence of adverse medication events in the perioperative setting | 6 months
  Number of adverse medication events / number of medications administered
Preventability of medication errors and adverse medication events | 6 months
  Four-point Likert scale for preventability: definitely preventable, probably preventable, probably not preventable, and definitely not preventability
Severity of harm (or potential harm) associated with both medication errors and adverse medication events in the perioperative setting | 6 months
  Four-point Likert scale for severity:
  Fatal
  Life-threatening: The event has the potential to cause symptoms that if not treated would put the patient at risk of death.
  Serious: The event has the potential to cause symptoms that are associated with a serious level of harm that is not high enough to be life-threatening.
  Significant: The event has the potential to cause symptoms that while harmful to the patient pose little or no threat to the patient's function.

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Nanji, M.D., M.P.H., Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Nanji KC, Patel A, Shaikh S, Seger DL, Bates DW. Evaluation of Perioperative Medication Errors and Adverse Drug Events. Anesthesiology. 2016 Jan;124(1):25-34. doi: 10.1097/ALN.0000000000000904. PMID 26501385